CLINICAL TRIAL: NCT03991468
Title: Clinical Validation for Non-Inferiority of Primary Diagnosis by WSI Hamamatsu NanoZoomer S360MD Digital Slide Scanner System Compared to Conventional Determination by Light Microscope
Brief Title: Primary Diagnosis Study for Validation of Hamamatsu NanoZoomer S360MD Digital Slide Scanner System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamamatsu Photonics K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: HCT-P001
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Pathology
MeSH Terms: interventions — Diagnostic Imaging; Microscopy

STUDY DESIGN:
Intervention Model Description: Cases are assessed using both glass slide light microscopy and NanoZoomer digital whole slide imaging in a random order
Who Masked: Outcomes Assessor
Masking Description: Adjudicators are blinded to the imaging modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NanoZoomer Whole Slide Imaging (Experimental): All cases will be assessed via Whole Slide Imaging using the Hamamatsu NanoZoomer S360MD Digital Slide Scanner System to assess pathological characteristics of scanned slides.
  Interventions: Diagnostic Test: Whole Slide Imaging
- Glass Slide Light Microscopy (Active Comparator): All cases will be assessed via the use of traditional light microscopy to assess pathological characteristics of glass slides.
  Interventions: Diagnostic Test: Light Microscopy

INTERVENTIONS:
Diagnostic Test: Whole Slide Imaging — Scanning of a glass slide to create a digital image that can be viewed on a monitor
  Other Names: NanoZoomer Scanning & Imaging
  Arms: NanoZoomer Whole Slide Imaging
Diagnostic Test: Light Microscopy — Use of traditional light microscopy per institutional standard practice
  Arms: Glass Slide Light Microscopy

SUMMARY:
The primary objective of this study is to evaluate the safety and accuracy of the Hamamatsu WSI compared to those of the reference method (conventional light microscope (Glass)) under clinical use conditions as an aid for pathologists to view, review and diagnose digital images of surgical pathology slides.

The primary endpoint is the indicator of major discordance in primary diagnosis between ground truth case diagnosis and case diagnosis by each modality, WSI and Glass, separately.

ELIGIBILITY:
Inclusion Criteria:

* Cases originating from and that were diagnosed at that local site
* Cases are available in the site's archive
* Cases are at least 1 year old since accessioning
* Cases are selected because their primary diagnosis is consistent with the assigned target categories
* Cases have a set of slides representative of the primary diagnosis for which it has been selected

Slide selection for a given case must meet the following criteria:

* Slide is obtained by surgical pathology and prepared from FFPE human tissue
* Slides must be stained with H&E and accompanying special stains (histochemical and/or immunohistochemical)
* All special stains slides (histochemical and/or immunohistochemical) where the slide and stain is used for diagnosis, not prognosis.
* A chosen slide must demonstrate and be representative of the primary diagnosis; 1 slide selection may suffice for biopsy cases,
* For resection cases, a minimum of 5 slides must be selected, which represent the primary diagnosis. If represented with less than 5 slides, additional slides (primary, secondary, or benign slides) from same case may be used to fulfill minimum number
* Slide is intact, has correct size/thickness, good edges, undamaged coverslip, without pen markings that can't be removed, no air bubbles, tidy labels, and fulfills the quality checks per the general clinical practice

Exclusion Criteria:

* Case does not have relevant slides or if case information necessary for the study is missing
* Case is still active (less than 1 year old) at the local site
* Cases for which the control slides for immunohistochemistry and special stains are not available
* Two cases from same individual
* Gross-only cases that have no slides
* Cases that are frozen section, cytology or hematology or immunofluorescence specimens only
* Case where the only available set of slides have evidence only of secondary or no diagnoses and not the primary diagnosis for which the case is being screened.

Slides for a given case will be excluded if they meet the following criterion:

• Glass slide that is broken, has abnormal size/thickness, beveled edges, poor coverslip (cracks, waviness, scratches), is sticky, has many pen markings or dirt that cannot be removed, contains air bubbles and overhanging labels that can't be corrected, and if stain is severely faded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liron Pantanowitz, Principal Investigator — University of Pittsburgh Medical Center
Locations (4):
- United States (4):
  - Washington University, St Louis, Missouri
  - TriCore Reference Laboratories, Albuquerque, New Mexico
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cases were assessed using both glass slide light microscopy and digital whole slide imaging in a random sequence. Therefore, each case had 2 primary diagnoses in the study.
Groups:
- All Cases: All cases will be assessed via Whole Slide Imaging using the Hamamatsu NanoZoomer S360MD Digital Slide Scanner System to assess pathological characteristics of scanned slides and traditional light microscopy using glass slides. The order in which each modality is used will be randomly assigned.
Period: Overall Study
Arm/Group | All Cases
Started | 2000
Glass Slide Light Microscopy | 2000
NanoZoomer Whole Slide Imaging | 2000
Completed | 2000
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Cases: All cases were assessed via Whole Slide Imaging using the Hamamatsu NanoZoomer S360MD Digital Slide Scanner System to assess pathological characteristics of scanned slides and traditional light microscopy using glass slides. The order in which each modality is used was randomly assigned.
Arm/Group | All Cases
Number analyzed (Participants) | 2000
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1046
  Male | 954
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2000

OUTCOME MEASURES:

1. Primary Outcome: Major Discordance Rate
Description: Indpendent reads by four Reading Pathologists (RPs) of both imaging modalitites (8 reads/case) were compared to the original diagnosis ("ground truth" or GT) by an independent adjudication process. This resulted in one of four adjudication outcomes for each read: "Match" (read = GT), "Minor" (minor discordance between read & GT), "Major" (major discordance between read & GT), or "Deferred" (read deferred by RP and excluded from the primary endpoint analysis). The outcome measure was the rate at which major discordances occurred for each modality.
Time Frame: 1 day
Population: Two modalities (glass & WSI) are read by 4 reading pathologists at each site for a total of 16,000 reads. Any reads deferred by a reading pathologist are excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of Major Discordances
Units Other Than Participants: Reads
Groups:
- NanoZoomer Whole Slide Imaging: Whole Slide Imaging using the Hamamatsu NanoZoomer S360MD Digital Slide Scanner System to assess pathological characteristics of scanned slides
  Whole Slide Imaging: Scanning of a glass slide to create a digital image that can be viewed on a monitor
- Glass Slide Light Microscopy: Use of a traditional light microscope to assess pathological characteristics of glass slides
  Light Microscopy: Use of traditional light microscopy per institutional standard practice
Arm/Group | NanoZoomer Whole Slide Imaging | Glass Slide Light Microscopy
Number analyzed (Participants) | 2000 | 2000
Number analyzed (Reads) | 7997 | 7998
Percentage of Major Discordances | 3.5 [2.6 to 4.7] | 3.1 [2.2 to 4.2]
Statistical Analysis 1: Comparison: NanoZoomer Whole Slide Imaging vs Glass Slide Light Microscopy; Test type: Non-Inferiority — A Mixed Model Repeated Measures logistic regression was used to prove WSI major discordance (MD) rate non-inferior to Glass MD rate. A two-sided 95% CI for the difference in MD rate was constructed. If the upper bound of the 95% CI was less than the non-inferiority margin of 4%, then WSI would be considered non-inferior to Glass, assuming power = 0.9 and alpha = 0.05 a sample size of 2000 was calculated to be sufficient to prove non-inferiority; Mixed Models Analysis; Dependent var = major discordance status (yes/no); independent var = modality (WSI/Glass) as a fixed effect & site, reader, & case as random effects; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 1.0]

ADVERSE EVENTS:
Time Frame: Because there was no patient involvement in the study and no impact on patient diagnoses, there were no safety endpoints for the study
Description: Because there was no patient involvement in the study and no impact on patient diagnoses, there were no safety endpoints for the study. Therefore no adverse event assessment or monitoring took place.
Arm/Group | All Cases
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03991468/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03991468/SAP_002.pdf